CLINICAL TRIAL: NCT03481907
Title: Topical Collagen Powder as a Wound Healing Adjuvant for Acute Full-thickness Punch Biopsy-induced Human Wounds: a Pilot Study
Brief Title: Topical Collagen Powder for Healing of Acute Full-thickness Wounds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adam Friedman (Other)
Collaborators: CPN Biosciences (Industry)
Responsible Party: Sponsor-Investigator, Adam Friedman, Principal Investigator, George Washington University
Organization: George Washington University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 26552436
Record Dates: First submitted 2018-03-15; First posted 2018-03-29 (Actual); Results first posted 2023-03-28 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Wound of Skin; Wound Heal
Keywords: collagen powder; punch biopsy wound

STUDY DESIGN:
Intervention Model Description: This is a self-controlled trial in which subjects will receive punch biopsies at sites on each leg, and will receive a different treatment on each of the 2 sites.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Internalized Control (Other): Subjects will receive 2 punch biopsy created wounds, one on each thigh, which will be addressed with primary closure with sutures or will be treated with Nuvagen collagen powder at time of wounding and daily thereafter. Suture(s) will be removed in 2 weeks. At week four, the wounded site will be biopsied again for tissue collection/evaluation, and treated with primary closure again. Suture(s) will be removed within to weeks. For those using collagen powder, the biopsy site will be biopsied again at week 4, and wound care will again be with NuvagenTM collagen powder until closure.
  Interventions: Device: Nuvagen Collagen Powder

INTERVENTIONS:
Device: Nuvagen Collagen Powder — Daily application of Nuvagen collagen powder for 2 to 4 weeks following wounding

SUMMARY:
We have designed a pilot study to investigate the effect and potential utility of topical NuvagenTM (collagen powder) on the rate and quality of wound healing in healthy volunteers using the punch biopsy method. After inducing an acute full-thickness wound, the rate of complete healing of a wound treated with topical NuvagenTM (collagen powder) will be compared to the rate of complete healing of a wound treated with primary closure with sutures, the current gold standard. Qualification and semi-quantification of histologic and immunohistochemical markers will be used to assess the maturity and structural stability of the wound bed. Positive findings would suggest that NuvagenTM (collagen powder) may be capable of stimulating the healing of acute wounds in a similar or even superior manner to primary closure, suggesting collagen powder may be used in place of sutures, and encouraging further studies to characterize its therapeutic potential in dermatologic surgery.

DETAILED DESCRIPTION:
Each patient received a single 4mm punch biopsy on each anterior thigh to provide for internalized controls. One wound was managed with PC, while the other was treated with daily topical collagen powder for up to four weeks. Prior to each biopsy, the areas were cleansed with an alcohol swab and anesthetized using 1 mL of 2% lidocaine with epinephrine. An Integra Miltex 4.0 mm Standard Biopsy Punch instrument was used to create full-thickness wounds and pressure was applied with gauze until hemostasis occurred.

Up to one gram of topical type 1, 100% bovine collagen powder (NuvagenTM, CPN Biosciences, Inc., Largo, FL) was placed on one wound before covering it with a non-adherent sterile dressing. The other wound underwent PC with two epidermal sutures (Ethilon Nylon Sutures, Ethicon, Somerville, NJ) and was similarly covered with a sterile dressing. At the four week follow-up, wounds were re-biopsied following the same procedures.

For home treatment, patients were provided with collagen powder in one-gram containers and dressings along with the following instructions: 1) Irrigate the wound with tap water or saline solution, 2) Dry the wound with gently with dry gauze, 3) Apply up to one gram of collagen powder to the wound, and 4) Apply a sterile dressing. Assistance from a caregiver was permitted as needed. This procedure was repeated daily for four weeks after the first biopsy and until wound closure after the second biopsy. For wounds closed primarily, patients were instructed to apply petroleum jelly before covering the wounds with sterile dressings.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient, male or female subjects of any race, 18-75 years of age
* Able to understand the requirements of the study and understand and sign Informed Consent/HIPAA Authorization forms
* Patients willing to refrain from using topical medications to punch biopsy sites
* Patients who are willing to follow protocol instructions and return for follow-up visits

Exclusion Criteria:

* Patients that have any medical or skin condition that could impair wound healing
* Patients that have used systemic medications that suppress the immune system within 5 half-lives (if known), or 2 months of enrollment (i.e. corticosteroids)
* Patients that have applied topical steroids to the thigh(s) in the 2 weeks prior to enrollment
* Patients that are currently participating in an investigational study of a drug or device or have participated within 4 weeks of enrollment
* Patients that in the opinion of the investigator demonstrate evidence of unwillingness or inability to follow instructions or to complete the study
* Patients currently using systemic antimicrobials
* Patients with a history of diabetes mellitus
* Patients with a history of bleeding disorders or concomitant treatment with aspirin or anticoagulants (including heparin, low molecular weight heparin, warfarin, fondaparinux, or rivaroxaban)
* Patients with a history of keloids or hypertrophic scars
* Patients with other conditions considered by the investigator to be reasons for disqualification that may jeopardize subject safety or interfere with the objectives of the trial (e.g., acute illness or exacerbation of chronic illness)
* Patients with a known allergy or sensitivity to any component of the test medication (including bovine and/or collagen products) or local anesthetic agent used
* Current or previous users of tobacco products
* Recent alcohol or drug abuse is evident
* Pregnant females or nursing mothers. Eligible women of reproductive age will be required to have a negative urine pregnancy test at screening. They will also be required to be on at least 1 reliable form of effective birth control [examples: barrier method (condoms, diaphragm), oral, injectable, implant birth control or abstinence] during the course of this study and 30 days following the last treatment period.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2018-10-18 (Actual); Study Completion 2018-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Friedman, MD, Principal Investigator — GW School of Medicine and Health Sciences
Locations (1):
- George Washington Medical Faculty Associates, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Yes
The results are published in Journal of Dermatology and Drugs
Supporting Information: Study Protocol, SAP
Time Frame: The data will be available for public reference after JAN 29 2018
Access Criteria: Journal of Dermatology and Drugs online access
URL: https://pubmed.ncbi.nlm.nih.gov/31334925/

REFERENCES:
- [Derived] Qureshi A, Murphy E, Milando R, Rengifo-Pardo M, Clayton C, Friedman A. A Head-to-Head Comparison of Topical Collagen Powder to Primary Closure for Acute Full-Thickness Punch Biopsy-Induced Human Wounds: An Internally Controlled Pilot Study. J Drugs Dermatol. 2019 Jul 1;18(7):667-673. PMID 31334925

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eight healthy volunteers 18 to 75 years old were enrolled after Informed consent form was signed for this study
Pre-assignment Details: Healthy patients 18 -75 years included. Patients with impaired wound healing, systemic immunosuppressants use within 2 months, steroid application to the thighs 2 weeks, participation in investigational trials in less than 4weeks , systemic antibiotics use , History of Diabetes Mellitus, bleeding disorders, keloids, hypertrophic scarring, allergy to collagen powders, current or past history of tobacco, alcohol or other illicit drug us and pregnant or nursing females were excluded.
Units Other Than Participants: left and right thighs of each subject
Groups:
- All Study Participants: All Subjects will receive 2 punch biopsy created wounds, one on each thigh to provide internalized controls, one thigh wound either left or right randomly which will be treated with primary closure( sutures) other thigh will be treated with Nuvagen collagen powder covered with sterile dressing at time of biopsy and daily thereafter for 4 weeks. Suture(s) will be removed in 2 weeks. Results are read to assess healing with wound size. At week four, both the wounded sites will be biopsied again to assess pathology results for healing tissue evaluation, and treated with primary closure again. Suture(s) will be removed within two weeks.
Period: Overall Study
Arm/Group | All Study Participants
Started | 8; 16 left and right thighs of each subject
Two Biopsies One on Each Thigh at Day 0 With Photo IHC and Histopathological Processing | 8; 16 left and right thighs of each subject
One Biopsy Wound Managed With Primary Closure | 8; 8 left and right thighs of each subject
Other One Biopsy Wound Managed With Topical Collagen Powder for 4 Weeks | 8; 8 left and right thighs of each subject
Photos of Both Wounds Were Taken at Week 46 With a Ruler in the Frame for Size Calibration | 8; 16 left and right thighs of each subject
Immunohistochemistry Done at 4 Weeks to Determine Collagen Content by Performing a Second Biopsy | 8; 16 left and right thighs of each subject
Completed | 8; 16 left and right thighs of each subject
Not Completed | 0; 0 left and right thighs of each subject

BASELINE CHARACTERISTICS:
Population: Eight healthy volunteers 18-75 years old were enrolled after providing informed consent. Exclusion criteria included chronic diseases, tobacco use, pregnancy, and other factors that could affect wound healing. Patients with a history of bleeding disorders, keloids, or hypertrophic scars were excluded to minimize adverse effects
Groups:
- All Participants: Biopsy of one anterior thigh of all patients followed by wound care with Primary Closure. Biopsy of other anterior thigh in all patients followed by wound care with Collagen powder
Arm/Group | All Participants
Number analyzed (Participants) | 8
Age, Continuous [Mean (Full Range); unit: years] — 8 patients from the GWU ambulatory clinics were consented for voluntary participation
  years | 37 [23 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8
Fitz-Patrick Skin type [Count of Participants; unit: Participants] — Skin type features Tanning I Pale white skin, light eyes and hair Always burns, does not tan II Fair skin, blue eyes Burns easily, tans poorly III Darker white skin Tans after initial burn IV Light brown skin Burns minimally, tans easily V Brown skin Rarely burns, tans darkly easily VI Dark brown or black skin Never burns, always tans darkly
  Participants
    Type I | 1
    Type II | 3
    Type III | 1
    Type III-IV | 2
    Type IV | 0
    Type V | 1
    Type VI | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Wound Diameter
Description: Change in wound diameter will be assessed digitally from photographs of the wounds obtained at several distinct time points, both at the time of wounding and afterwards. The diameter of the biopsy wound is measured to reflect a change from baseline in wound size day 0 and again at week 4.
Time Frame: 4 weeks after first biopsy
Population: 8 voluntary out patients were selected between ages 18 and 75, 2 female subjects. There was one patient with Fitzpatrick Skin type (FST) I, Three were FST II, one FST III, tow, FST III/IV, and one FST V.
Measure: Mean (90% Confidence Interval); unit: Centimeters
Groups:
- Primary Closure: All Subjects will receive a punch biopsy, on one thigh, which will be closed with primary closure suture(s) , removed in 2 weeks. At week four, the wounded site closure will be measured by its diameter after which the site will be biopsied again for tissue collection to evaluate collagen content by pathology and immunohistochemistry (IHC), and treated with primary closure. Suture(s) will be removed in 2 weeks.
- Collagen Powder: All subjects will receive biopsy on the other thigh, and wound care will again be with NuvagenTM collagen powder. Biopsy wound treated with daily topical collagen powder for up to four weeks . At week four, the wounded site closure will be measured by its diameter after which the site will be biopsied again for tissue collection to evaluate collagen content by pathology and immunohistochemistry (IHC), and treated with primary closure. Suture(s) will be removed in 2 weeks.
Arm/Group | Primary Closure | Collagen Powder
Number analyzed (Participants) | 8 | 8
Centimeters | 95.94 [91.81 to 99.47] | 95.94 [92.41 to 99.47]

2. Other Pre Specified Outcome: Collagen Staining in Histopathology
Description: histopathological processing was performed by HistoWiz, Inc. (Brooklyn, NY) on one baseline sample and both four-week samples, including hematoxylin and eosin (H&E), CD31 (platelet-derived endothelial cell adhesion molecule-1), and Masson trichrome staining. H&E staining was used to examine the quality of the epidermis and colla- gen bundles as well as to observe the amount of inflammatory granulation tissue.
Time Frame: at 4 weeks after first biopsy
Population: as for outcome 1
Measure: Mean (90% Confidence Interval); unit: percentage of Masson trichrome staining
Groups:
- Primary Closure: Subjects will receive 2 punch biopsy created wounds, one on each thigh, which will be addressed with primary closure with sutures or will be treated with Nuvagen collagen powder at time of wounding and daily thereafter. Suture(s) will be removed in 2 weeks. At week four, the wounded site will be biopsied again for tissue collection/evaluation, and treated with primary closure again. Suture(s) will be removed within to weeks. For those using collagen powder, the biopsy site will be biopsied again at week 4, and wound care will again be with NuvagenTM collagen powder until closure.
  Nuvagen Collagen Powder: Daily application of Nuvagen collagen powder for 2 to 4 weeks following wounding
Arm/Group | Primary Closure | Collagen Powder
Number analyzed (Participants) | 8 | 8
percentage of Masson trichrome staining | 125.8 [118.49 to 133.11] | 173.40 [164.07 to 182.73]

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: No difference in definition of Adverse reaction than as defined by clinicaltrials.gov.
  The procedure is a simple routine with very low risk to threat of adversity
Groups:
- Primary Closure: All subjects will receive punch biopsy on anterior one thigh and wound care is by primary closure with suture
- Collagen Powder: All subjects will receive punch biopsy on othe ranterior thigh and wound care is bycollagen powder and dressing
Arm/Group | Primary Closure | Collagen Powder
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8

LIMITATIONS AND CAVEATS:
Small sample size, absence of negative control

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-29): https://cdn.clinicaltrials.gov/large-docs/07/NCT03481907/Prot_SAP_004.pdf